CLINICAL TRIAL: NCT07011654
Title: Phase I/II Study of Naxitamab and Sacituzumab Govitecan in Patients With Metastatic Triple-negative Breast Cancer (TNBC)
Brief Title: Study of Naxitamab and Sacituzumab Govitecan in Patients With Metastatic Triple-negative Breast Cancer (TNBC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0438; NCI-2025-03798 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-05-30; First posted 2025-06-09 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan; naxitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with Naxitamab and Sacituzumab Govitecan IV Q3W (Experimental): Patients receive naxitamab IV on days 2, 4, and 6 of cycles 1-8 and sacituzumab govitecan IV days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab govitecan; Drug: Naxitamab

INTERVENTIONS:
Drug: Sacituzumab govitecan — Given by IV
Drug: Naxitamab — Given by IV

SUMMARY:
This phase I/II trial tests the safety, best dose, and effectiveness of naxitamab in combination with sacituzumab govitecan in treating patients with triple-negative breast cancer (TNBC) that has spread from where it first started (primary site) to other places in the body (metastatic).

DETAILED DESCRIPTION:
1. Primary Objectives

   * To determine the safety and tolerability and establish the maximum tolerated dose/recommended phase 2 dose (MTD/RP2D) of the combination of naxitamab and sacituzumab govitecan in participant s with metastatic TNBC.
   * To determine the objective response rate (ORR) of naxitamab in combination with sacituzumab govitecan per RECIST v1.1 criteria in participant s with metastatic TNBC at the MTD/RP2D.
2. Secondary Objectives

   * To determine the duration of response, progression-free survival, and overall survival for participant s with metastatic TNBC treated with the combination of naxitamab plus SG:
   * To identify GD2-related biomarkers of response and resistance to the combination of naxitamab and sacituzumab govitecan.
3. Exploratory/Correlative Objectives • Investigate potential resistance mechanisms to naxitamab and develop a pre-clinical rationale for future therapeutic strategies.

ELIGIBILITY:
Inclusion criteria

* Male and female participants aged 18 years or older and able to understand and give written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 (for the phase I portion of the study) and ECOG performance status of 0-2 (for the phase II portion of the study)
* Life expectancy of at least 3 months
* Histologically confirmed metastatic TNBC. (Estrogen receptor [ER] ≤10%; Progesterone receptor [PgR] ≤10%, HER2-negative as per ASCO/CAP guidelines)
* Willingness to provide archival tumor tissue for correlative studies associated with this trial.
* Received at least 1 prior line of systemic chemotherapy for metastatic TNBC and/or meet criteria to receive sacituzumab govitecan as standard of care
* Measurable disease by CT or MRI as per RECIST Version 1.1 criteria
* Adequate organ and marrow function as defined below:

  2. Exclusion Criteria Participants who meet any of the following exclusion criteria are not eligible to be enrolled in this study.
* Positive serum pregnancy test or women who are lactating.
* Known or severe (≥ Grade 3) hypersensitivity or allergy to naxitamab and/or sacituzumab govitecan, their metabolites, or formulation excipient.
* Grade 3 or greater peripheral neuropathy
* Have previously received treatment with an anti-GD2 antibody
* Prior treatment with TROP2-targeting antibody drug conjugates in the metastatic setting. Participant s who have received TROP2-targeting antibody drug conjugates in the neoadjuvant setting or adjuvant setting are eligible if at least 6 months have elapsed since the last dose of TROP2-targeting antibody drug conjugate.
* Have an active second malignancy. Participant s with a history of active cancer for 3 years prior to enrollment, or participant s with surgically cured tumors with low risk of recurrence (eg, nonmelanoma skin cancer, histologically confirmed complete excision of carcinoma in situ, or similar) are allowed to enroll.
* Have known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Have undergone an allogenic tissue or solid organ transplant.
* Uncontrolled hypertension, defined as a consistently elevated systolic blood pressure of >160 mmHg despite optimal medical management
* Clinically significant cardiac disease
* Inadequate pulmonary function
* Active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrollment.
* Uncontrolled seizure disorders despite anticonvulsant therapy (defined as a seizure event within 3 months prior to enrollment)
* Active serious infection requiring systemic antimicrobial therapy.
* Participants positive for HIV-1 or 2 with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
* Have active hepatitis B or C infection
* Has a diagnosis of immunodeficiency or receiving systemic corticosteroid therapy (higher than physiologic doses) ≥ 10 mg of prednisone per day or equivalent] or any other form of immunosuppressive therapy within 14 days of initiation of study treatment.
* Has received prior radiotherapy within 1 weeks of start of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Clinton Yam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org